CLINICAL TRIAL: NCT04328207
Title: Using Telemedicine to Prevent Blindness in an At-risk Rural Alabama Population
Brief Title: Providing Financial Incentives to Improve Adherence to Referral Eye Care Visits
Acronym: AL-SIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Owsley, Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRB-300004921; 1U01DP006441-01-00 (Other: Centers for Disease Control); 1U01DP006441-01 (NIH)
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Glaucoma; Diabetic Retinopathy; Refractive Errors; Cataract; Behavior, Health
Keywords: telemedicine; teleophthalmology; telehealth; teleglaucoma; financial incentives
MeSH Terms: conditions — Glaucoma; Diabetic Retinopathy; Refractive Errors; Cataract; Health Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: In the first half of enrollment in the program there will be no financial incentive offered to any patients. In the second half of enrollment, all patients needing referral will be notified that they will receive a payment upon the completion of their referral visit.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators are masked as to which group the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No financial incentive (Other): This group will receive standard of care eye health education alone and no financial incentive for completing a referral visit.
  Interventions: Other: No Financial Incentive
- Financial incentive (Experimental): This group will receive a financial incentive once the referral visit is completed (if one was required) as well as eye health education.
  Interventions: Behavioral: Financial Incentive

INTERVENTIONS:
Other: No Financial Incentive — Standard of care eye health education
  Other Names: Standard of Care
  Arms: No financial incentive
Behavioral: Financial Incentive — Patients who are referred for an in-person follow-up exam will receive a financial incentive once the referral visit is completed.
  Arms: Financial incentive

SUMMARY:
Glaucoma is a blinding eye disease increasingly common in older adults, particularly in African Americans, and often diagnosed late in the disease course. It is essential to develop novel health care models, utilizing telemedicine, to improve the ability to detect glaucoma at an earlier stage, and to provide a platform to manage this disease in community-based clinics so that further vision loss is prevented. Our goal is to improve the quality and accessibility of glaucoma detection and management among a vulnerable and at-risk segment of our population.

DETAILED DESCRIPTION:
The number of primary open angle glaucoma (POAG) cases will increase by 250% by 2050, directly affecting over 7 million lives. These numbers are specifically for POAG and do not include the many who are monitored and treated for elevated intraocular pressure or for glaucoma suspect status, which along with POAG can all be considered glaucoma associated diseases (GAD). Development of high-quality, accessible, and cost-effective strategies for eye care for these individuals is of critical importance. POAG is at least 4-5 times higher in African Americans, progresses more rapidly and appears about 10 years earlier as compared to those of European descent. This research plan seeks to implement and evaluate a telemedicine-based detection and management strategy for GAD and other eye diseases in patients seen at Federally Qualified Health Centers (FQHC's) located in the rural Alabama Black Belt Region. This region is characterized by one of the highest concentrations of African Americans in the US; high poverty, unemployment, and uninsured rates; inadequate educational systems, transportation and community resources; few optometrists who largely practice in retail settings; and no ophthalmologists specializing in glaucoma. The investigators have developed and tested a novel multimodal telemedicine approach in a prior Centers for Disease Control and Prevention (CDC) funded Eye Care Quality and Accessibility Improvement in the Community (EQUALITY) study that used comprehensive remote optic nerve assessment (RONA). This proposal will employ a modification of the EQUALITY approach using portable measurement of visual function and optic nerve and retinal structure that are more applicable to rural locations with limited resources. The investigators will also identify and evaluate remediation strategies for the barriers to patient adherence with referral and follow-up appointments by comparing the effectiveness of financial incentives along with a validated patient education program versus a validated patient education program alone. Using this program within FQHC's will enable expansion nationwide into rural and urban underserved locations as these centers provide primary health care services in underserved areas and treat more than 27 million people yearly at over 12,000 sites.

ELIGIBILITY:
Inclusion Criteria:

* African American or Hispanic ≥40 years
* Non-Hispanic white ≥50 years
* Anyone ≥ 18 years with diabetes
* Anyone ≥ 18 years with a glaucoma associated diagnosis
* Anyone ≥ 18 years with a family history of glaucoma
* All enrollees must be able to speak and understand English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Girkin, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined at a later point.

REFERENCES:
- [Derived] Rhodes LA, Register S, Asif I, McGwin G Jr, Saaddine J, Nghiem VTH, Owsley C, Girkin CA. Alabama Screening and Intervention for Glaucoma and Eye Health Through Telemedicine (AL-SIGHT): Study Design and Methodology. J Glaucoma. 2021 May 1;30(5):371-379. doi: 10.1097/IJG.0000000000001794. PMID 33492893
- See also: Website describing the research program as well as two other research programs funded by the same mechanism. — https://sightstudies.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Financial Incentive | Financial Incentive
Started | 499 | 401
Completed | 499 | 401
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Financial Incentive | Financial Incentive | Total
Number analyzed (Participants) | 499 | 401 | 900
Age, Categorical [Count of Participants; unit: Participants] — From electronic medical record
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 272 | 200 | 472
    >=65 years | 227 | 201 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.49 (13.50) | 59.58 (11.99) | 58.97 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 322 | 258 | 580
  Male | 177 | 143 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 496 | 397 | 893
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 228 | 142 | 370
  White | 257 | 250 | 507
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 9 | 23
Region of Enrollment [Number; unit: participants]
  United States | 499 | 401 | 900

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Adhere to Referral Appointment
Description: The percentage of patients who adhere to attending their referral appointments who received a financial incentive and eye health education will be compared with the percentage of patients who adhere to attending their referral appointments who received standard of care eye health education alone and no financial incentive for completing a referral visit.
Time Frame: The time frame will be whether they attended the referral appointment between the screening date until 6 months after the screening date.
Measure: Count of Participants; unit: Participants
Arm/Group | No Financial Incentive | Financial Incentive
Number analyzed (Participants) | 499 | 401
Participants | 80 | 92

ADVERSE EVENTS:
Time Frame: 24 months
Description: The definition of an adverse event is as defined by clinicaltrials.gov.
Arm/Group | No Financial Incentive | Financial Incentive
All-Cause Mortality (participants affected / at risk) | 0/499 | 0/401
Serious Adverse Events (participants affected / at risk) | 0/499 | 0/401
Other Adverse Events (participants affected / at risk) | 0/499 | 0/401

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04328207/Prot_SAP_000.pdf